CLINICAL TRIAL: NCT03472664
Title: Brain Energy for Amyloid Transformation in AD (BEAT-AD) Study
Brief Title: Brain Energy for Amyloid Transformation in Alzheimer's Disease Study
Acronym: BEAT-AD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00049474; 1R01AG055122-01 (NIH)
Record Dates: First submitted 2018-03-12; First posted 2018-03-21 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-04

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment
Keywords: Memory; Diet; ketogenic
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Adults with amnestic mild cognitive impairment will be randomized on a 1:1 schedule to receive either a 4-month Modified Mediterranean Ketogenic Diet or American Heart Association Diet intervention. Diet interventions will be equicaloric with participants' normal diets. Personalized nutritional guidance and menus will be provided, and compliance will be assessed by a registered dietitian. Amyloid positron emission tomography (PET) will be conducted at baseline. Blood collection and cognitive assessment will be conducted at baseline and after 2 and 4 months of diet. Lumbar puncture (LP) and MRI will be conducted at baseline and following the intervention for all participants.
Who Masked: Investigator, Outcomes Assessor
Masking Description: It is not possible for participants and the dietitian to be blinded to the study diet.
  Study personnel involved in performing cognitive testing or other outcome procedures or data analysis will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified Mediterranean Ketogenic Diet (Experimental): The MMKD is a low carbohydrate/high fat diet aimed at inducing ketosis, as the experimental diet in the proposed study. Participants on the MMKD will keep their daily carbohydrate consumption below 20 grams per day throughout the 4 month intervention.The MMKD group will be supplied with extra virgin olive oil during their in person visits to use as a source of fat in their diet, and will be encouraged to eat plentiful fish, lean meats, and nutrient rich foods that meet the requirement of <20 grams total carbohydrates per day.
  Participants will receive a daily multivitamin (Centrum Silver) over the course of the study and instructed to take 1 tablet each day while on the diet.
  Interventions: Other: low carbohydrate/high fat diet
- American Heart Association Diet (Experimental): The American Heart Association Diet (AHAD), is a low fat/high carbohydrate diet (<40 grams/day) will be used as the control diet. Participants on the AHAD will be encouraged to limit their amount of fat intake to <40 grams/day, while eating plentiful fruits, vegetables, and carbohydrates containing adequate fiber. Participants will receive the same daily multivitamin supplement (Centrum Silver) over the course of the study and instructed to take 1 tablet each day while on the diet.
  Interventions: Other: low fat/high carbohydrate diet

INTERVENTIONS:
Other: low carbohydrate/high fat diet — Modified Mediterranean-Ketogenic Diet is a low carbohydrate/high fat diet.
  Arms: Modified Mediterranean Ketogenic Diet
Other: low fat/high carbohydrate diet — American Heart Association Diet is a low fat/high carbohydrate diet.
  Arms: American Heart Association Diet

SUMMARY:
The Brain Energy for Amyloid Transformation in AD (Alzheimer's disease) or BEAT-AD study will compare the effects of a ketogenic low-carbohydrate diet and a low-fat diet in adults with mild cognitive impairment. The data collected will help determine whether diet interventions induce changes in cognitive function, cerebral blood flow, and levels of certain proteins and hormones in body fluids.

The study will include volunteers who have mild cognitive impairment, who will be randomly assigned to receive either a ketogenic low-carbohydrate diet or a low-fat diet for 16-weeks, with follow-up assessment 8 weeks after diet completion. Study measures, clinic visits and phone sessions will occur at baseline and throughout the 24-week study.

Participant will follow either a low-carbohydrate or low-fat diet that will be individually planned with help from a study dietitian. After completing the study diet for 16 weeks, participants will resume their normal diet. The final visits will occur at week 24 (8 weeks after the completing the diet). At the end of the 24-week study, participants will be given the opportunity to meet with the study dietitian for education and assistance with planning a healthy diet.

DETAILED DESCRIPTION:
This study will examine the effects of a 4-month Modified Mediterranean-Ketogenic Diet compared with an American Heart Association Diet (AHAD - a regimen that has been shown to reduce the risk for cardiovascular disease). We will investigate diet effects on AD biomarkers, on cognition, and on neuroimaging measures of blood flow. Our study will extend previous findings in several important ways by: 1) using a Modified Mediterranean-Ketogenic Diet rather than a traditional Ketogenic Diet, which has the potential for greater long-term compliance and health benefits; 2) increasing the sample size and duration of the diet intervention; 3) examining potential mechanisms of diet effects that may result in new biomarkers and therapeutic targets; and 4) examining key treatment response variables such as Apolipoprotein E (ApoE) genotype, amyloid positivity and metabolic status that could inform precision medicine approaches to dietary prescription.

Adults with amnestic mild cognitive impairment (MCI) will be randomized on a 1:1 schedule to receive either a 4-month Modified Mediterranean-Ketogenic Diet (MMKD) or American Heart Association Diet (AHAD) intervention. Diet interventions will be equicaloric with participants' normal diets. Personalized nutritional guidance and menus will be provided, and compliance will be assessed by a registered dietitian. The principal investigator will be responsible for the overall monitoring of the data and safety of study participants, with assistance by members of the study staff, and the Data and Safety Monitoring Board (DSMB), which will be responsible for monitoring the safety of research participants.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of amnestic mild cognitive impairment
* An informant (study partner) able to provide collateral information on the participant
* Stable medical condition (generally 3 months prior to screening visit) at the discretion of study physician
* Stable on medications (generally 4 weeks prior to screening visit) at the discretion of study physician
* Able to complete baseline assessments

Exclusion Criteria:

* Diagnosis of neurodegenerative illness (except for MCI);
* History of a clinically significant stroke
* Current evidence or history in past year of focal brain lesion, head injury with loss of consciousness or DSM-IV criteria for any major psychiatric disorder including psychosis, major depression, bipolar disorder, alcohol or substance abuse
* Sensory impairment (i.e.: visual or auditory) that would preclude the participant from participating in the protocol
* Diabetes that requires current use of diabetes medications
* Clinically significant elevations in liver function tests
* Active neoplastic disease (stable prostate cancer and non-melanoma skin cancer is permissible)
* History of epilepsy or seizure within past year
* Contraindications for MRI (claustrophobia, craniofacial metal implants, pacemakers)
* Significant medical illness or organ failure, such as uncontrolled hypertension or cardiovascular disease, chronic obstructive pulmonary disease, liver disease, or kidney disease

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-07-16 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Cerebrospinal Fluid (CSF) Abeta42 | 16 Weeks
  CSF Aβ42 is a a key AD biomarker that reflects pathological aggregation of amyloid in the brain.

SECONDARY OUTCOMES:
CSF abeta42/ptau ratio | 16 Weeks
  The ratio of CSF Aβ42 to tau is a key AD biomarker that reflects an integrated value of amyloid and tau pathology in the brain.
Preclinical Alzheimer Cognitive Composite (PACC) | 16 Weeks
  The PACC consists of Free and Cued Selective Reminding Test - Total Recall, Logical Memory IIa - Delayed Paragraph Recall, Digit Symbol Substitution Test, MMSE - Total Score and Category Fluency.
  Although the PACC was designed for use with preclinical AD, it is reasonable to assume it will also be sensitive in aMCI, as all PACC components are frequently used in aMCI studies. According to PACC developer, Reisa Sperling, MD, it is a useful indicator of cognitive change in aMCI in the Harvard Aging Brain Study (personal communication). Further, we observed significant improvement in our cognitive test composite that includes 2 PACC components following the MMKD.
Cerebral Blood Flow Measure with Arterial Spin Labeling (ASL) MRI | 16 Weeks
  Cerebral blood flow will be measured with pseudo continuous ASL MRI, and voxel based analyses will be conducted to determine diet-induced changes and their relationship to cognitive and biomarker outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Craft, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Medical Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Data sharing will follow guidelines and timeline recommended by the National Institute on Aging.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will become available one year after completion of the study and remain available indefinitely.
Access Criteria: Consultation with the study team to verify purpose of data sharing request, and collaborative involvement of study team if appropriate.